CLINICAL TRIAL: NCT03345628
Title: Feasibility Study to Determine Ability to Recruit and Assess Patients for a Neurodevelopment Follow-up Study in Pediatric Intensive Care
Brief Title: Feasibility Study for Neurodevelopment Follow-up Study in PICU
Acronym: PICUFUN
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Davinia Withington, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: PICU FUN 2018-3310
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Bronchiolitis Acute; Pneumonia
Keywords: sedation; critical care; infant; neurodevelopment
MeSH Terms: conditions — Pneumonia | interventions — Hypnotics and Sedatives

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sedated: infants requiring intubation and ventilation who received sedatives for at least 3 days
  Interventions: Drug: Sedatives
- non-sedated: infants who received respiratory support by non-invasive ventilation and were not sedated

INTERVENTIONS:
Drug: Sedatives — sedated group received sedative drugs to tolerated intubation and ventilation
  Other Names: sedation
  Groups: sedated

SUMMARY:
There is a large and growing body of animal evidence demonstrating neuroapoptosis and neurodevelopmental abnormalities after exposure to anesthetic agents. This has prompted an FDA warning concerning use of anesthetics and sedatives in children under 3 years of age. There has been very little investigation of the neurodevelopment effects of prolonged sedation in previously healthy infants in Paediatric Intensive Care. This feasibility study will recruit previously healthy infants who required respiratory support with or without sedation at up to 1 year of age and assess neurodevelopmental outcomes at 6 years of age.

DETAILED DESCRIPTION:
The majority of human cohort investigations of neurotoxicity have studied general anesthesia for surgery. However, many animal studies have involved exposure to agents for significantly longer than the average duration of a general anesthetic in infants, some even for 24 hours (8).This is closer in exposure characteristics to prolonged sedation in PICU: days as compared to a few hours. However, although sedation in the Pediatric Intensive Care Unit (PICU) may continue for several days, there are no studies of its effects on subsequent neurodevelopment in previously healthy young infants. The only intensive care studies thus far have examined high risk subgroups, including the EPIPAGE study (20) in premature newborns and studies of infants after congenital heart surgery. The latter studies have shown a small but significant association between cumulative benzodiazepine dose and Visual-Motor integration at 4 years of age (21), and an association between higher exposure to volatile anesthetic agents and lower cognitive scores on the Bailey Scales of Infant Development III at 12 months (22), respectively.

It is essential that Pediatric Intensivists start investigating the effect of our commonly used sedation protocols, which frequently include benzodiazepines, on our patients' neurodevelopment. The standard sedative regimen in use for many years at Montreal Children's PICU is midazolam infusion (benzodiazepine) plus opioid (commonly fentanyl or morphine) infusion. Other agents including ketamine may be added. This is not an easy field of study since we cannot randomize patients to receive sedation or not.

Therefore this programme of research aims to:

a) Identify a suitable group of PICU patients who were exposed to PICU sedation, along with a comparable group who were not exposed to sedation during their PICU admission who will act as controls; b) Assess the feasibility of recruiting these retrospectively identified patients and performing the requisite neurodevelopmental assessments around 6 years after PICU admission; c) Expand to a multicentre study, if feasibility is confirmed, to allow the recruitment of sufficient numbers of cases to determine if PICU sedation has a significant effect on long-term neurodevelopment; d) Investigate alternative sedation protocols and/or interventions to minimize the adverse effects on development.

1. The initial aim of this study programme has been achieved by means of a Chart Review completed in March 2017. We hypothesized that previously healthy infants requiring ventilation for an acute respiratory illness would divide into two groups depending on their respiratory management: intubation with sedation versus non-invasive ventilation without sedation, and that these infants, with a unifying pathological diagnosis, could act as cases and controls for an investigation of PICU sedation. In order to optimize the validity of our comparison, patients must be as similar as possible, therefore many exclusion criteria and also matching are required. The chart review has determined that the two described groups are similar in terms of severity of illness scores (Pediatric Risk of Mortality [PRISM] and Pediatric Logistic Organ Dysfunction [PELOD]) therefore making them suitable subjects for a follow-up study (23). This phase of the programme has been presented and discussed at Canadian Critical Care Trials Group (CCCTG) meetings and endorsed by CCCTG.
2. Having identified an appropriate group of patients, the next phase of the research programme is to perform a feasibility study to determine if our methodology will lead to adequate recruitment to move forward to a large multicentre study. This is the subject of this protocol.

The proposed methodology is similar to that used successfully in the PANDA study (16) where study participants were identified using billing records (hernia surgery at up to 36 months of age). Their records were checked for exclusion criteria based on age, gestational age at birth and general health. Parents were contacted and invited to participate. Further exclusions were based on more detailed medical history from the parents and the existence of a sibling within 3 years of the index child's age who had not had any anesthetic exposure and who was also healthy. Another general anesthesia study with similar methodology is currently analysing data (24). This group from the Mayo Clinic used population-based controls for anesthesia-exposed index cases identified from a previous cohort study (10). Our participant identification will also be retrospective, from medical records to identify sedation-exposed and non-exposed subjects from within the PICU population as described below.

Hypothesis: feasibility study Patients identified from the PICU admission records and Medical Records search can be suc-cessfully recruited and assessed by standard Neurodevelopmental testing 6 years after their admission.

Hypothesis: definitive study We hypothesize that benzodiazepines alone or with opioid infusion during mechanical ventilation of previously healthy infants with respiratory diagnoses would decrease Wechsler Preschool and Primary Scale of Intelligence III (WPPSI III) score at 6 yrs, compared to infants who were treated with non-invasive ventilation without sedation.

Aims for feasibility study

1. Identify patients from PICU database and from previous Chart Review Database (see below).
2. Recruit 20 patients each from the sedated/intubated/ventilated and non-sedated/non-invasive ventilation groups (total 40).
3. Perform pediatric and neurodevelopmental assessments on patients at 5 years 8 months to 7 years 4 months of age using a battery of tests with Wechsler Pediatric and Primary Infant scales of Development (IV) as the primary outcome.

Primary outcome Successful identification and recruitment of patients and performance of testing.

Secondary outcomes Performance of Wechsler Pediatric and Primary Infant scales of Development IV (WPPSI IV) and NEPSY-II™ tests at 5 years 8 months to 7 years 4 months .

Completion of Childhood Memory Score (CMS™) and Child Behaviour Checklist (CBCL)™ questionnaires Pediatric examination: incidence of neurological abnormalities including cerebral palsy, hearing or visual deficits, seizure disorder, Attention Deficit disorder, Autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* infants treated for bronchiolitis or pneumonia requiring respiratory support either intubation and IPPV needing sedation OR requiring non-invasive ventilation without sedation

Exclusion Criteria:

* prematurity less than 28 weeks, congenital heart disease, genetic or chromosomal anomalies, neurological disease, exposure to anesthesia in utero or prior to PICU admission, GA longer than 60 minutes or repeated PICU sedation since original admission.
* logistical exclusions: language other than English or French for which testing tools are available; geographical distance precluding return for testing appointment.

Max Age: 52 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PICU admissions for respiratory disease as specified in eligibility section recruited at 6 years of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Wechsler Pre-school and Primary Scale of Intelligence -IV | 6 years
  The Wechsler Preschool and Primary Scale of Intelligence consist of 14 subtests. They are designated as one of three types: core, supplemental, or optional. The core subtests are required for the computation of the Verbal, Performance, and Full Scale IQ. Quotient and Composite scores have a mean of 100 and a standard deviation of 15. Subtest scaled scores have a mean of 10 and a standard deviation of 3. A score of 90-109 is Average

SECONDARY OUTCOMES:
NEuroPSYchological Assessment (NEPSY) | 6 years
  The six functional domains below are made up of 32 subtests and four delayed tasks. These domains are theoretically, not statistically, derived. The subtests were designed to assess cognitive abilities related to disorders that are typically diagnosed in childhood and that are required for success in an academic environment.
Childhood Memory Scale (CMS™) | 6 years
  Pearson Clinical 5-8yrs record form. Assesses children's memory abilities. The CMS is administered to identify deficits in learning and memory. There are six core subtests and three supplemental subtests from which you can derive scaled scores (mean=10, SD=3). You may also derive eight Index Scores (mean 100, SD=15) from various combinations (summation) of subtest scaled scores: Visual Memory Immediate, Visual Memory Delayed, Verbal Memory Immediate, Verbal Memory Delayed, Verbal Memory Recognition, Attention/Concentration and Learning. Finally, Visual Memory Immediate, Visual Memory Delayed, Verbal Memory Immediate and Verbal Memory Delayed Indices can be summed to get a General Memory Score (mean 100, SD=15). A scaled score of 8-12 for the substests is average and a standard score of 90-110 forwppsi the indices is average.
Child Behaviour Checklist (CBCL)™ | 6 years
  widely used checklist assessing behaviours and emotional responses

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No